CLINICAL TRIAL: NCT02206906
Title: Investigation of Incentives to Promote Medication Adherence Among HIV-Infected Youth on Antiretroviral Therapy
Brief Title: Incentives to Promote Medication Adherence Among HIV-Infected Youth
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: INMED
Record Dates: First submitted 2014-07-30; First posted 2014-08-01 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2015-06

CONDITIONS: HIV
Keywords: Medication Adherence; Incentives; Real-time Medication Monitoring
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Participants: All participants who meet eligibility requirements and who consent to participation will use an incentive intervention model.
  Interventions: Behavioral: Incentive intervention model

INTERVENTIONS:
Behavioral: Incentive intervention model — All participants will receive a real-time electronic medication monitor to monitor daily pill-taking behavior. Participants with qualifying levels of adherence will receive a weekly incentive during the intervention period. At all clinic visits participants will participate in a lottery incentive to reinforce clinic attendance and negative STI screening tests.

SUMMARY:
Medication adherence is one of the most salient predictors of patient outcomes in the era following development of effective treatment for HIV infection. Evolving strategies to improve adherence, specifically incentive interventions and real-time medication monitoring, have shown some success in limited studies. Further investigation into incentive interventions for HIV-infected adolescents with poor medication adherence is necessary.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

* To describe the effects of a novel incentive intervention model on HIV-infected youths' patterns of antiretroviral medication adherence.

SECONDARY OBJECTIVES:

* To evaluate the feasibility of an outpatient incentive intervention model.
* To assess participant satisfaction with the incentive intervention model.
* To evaluate the effect of an outpatient incentive intervention model on targeted health behaviors (numbers of missed appointments and STI diagnoses).
* To measure the effect of the incentive intervention on HIV viral load and CD4+ count.
* To determine the overall and per patient cost of the incentive intervention model.
* To describe associations between adherence measures: real-time medication monitor data, pharmacy pill count, pharmacy prescription pick-up data, medication possession ratio, and self-report.

Upon enrollment, participants will receive education and a real-time medication monitor. Participants will be followed monthly in the clinic and will be prescribed thirty-day supplies of medication. During weeks 1-4 participants will establish a baseline with the real-time medication monitor. During weeks 5-28, participants will receive remote incentives based on their level of medication adherence as measured by the real-time medication monitor. Additional lottery-style incentives will occur at regular follow-up visits. No incentives will be applied during weeks 29-48. Participants will complete the protocol at the week 48 visit.

ELIGIBILITY:
Inclusion Criteria:

* ≥16 and ≤ 24 years old
* Documented diagnosis of HIV
* Adolescent is aware of his/her HIV diagnosis
* Adolescent understands either written or spoken English.
* Adolescent is willing and able to provide informed consent or assent.
* Adolescent has access to a phone and the internet at the time of enrollment.
* Adolescent meets the definition of inadequate ARV adherence, which is any of the following in the previous 12 months:

  * < 80% adherent to any ARV by pharmacy pill count
  * ≥ 7 days delay in scheduled ARV prescription pick-up
  * Detectable viral load after being on ARVs for at least 12 weeks

Exclusion Criteria:

* Adolescent has a documented diagnosis of mental retardation or a significant motor or sensory impairment that would preclude participation.
* Adolescent has a documented acute psychiatric illness, including suicidal ideation, homicidal ideation or active psychosis.
* Adolescent was diagnosed with HIV in the previous 6 months.
* Adolescent has a planned transition to alternative care setting prior to study completion (e.g. relocation, pregnancy or planned pregnancy, transition to adult care).
* Concurrent enrollment on a research study with an intervention targeted at increasing adherence to antiretroviral regimens.

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Youth with HIV who meet eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Percentage of dosages taken within 2 hours of prescribed time per month | Monthly through week 48
  Data collected by a real-time medication monitor that records pillbox opening times.
Pharmacy pill count | Monthly from 6 months prior to study start through week 48
  Pharmacy pill count data is collected at each participant encounter, approximately once per month.

SECONDARY OUTCOMES:
Feasibility - Accrual percentage | End of study (week 48)
  Number of people enrolled in study/number approached for enrollment.
Feasibility - Drop out rate | End of study (week 48)
  Number of people ending protocol early/ total enrollment
Feasibility - Participant reported device concerns | End of study (week 48)
  Problems with the Wisepill devices as spontaneously reported by participants or as assessed at routine follow-up.
Feasibility - Device replacement rate | End of study (week 48)
  Number of devices requiring replacement due to loss/theft/breakage
Feasibility - Contact failure rate | End of study (week 48)
  Number of failed attempts to contact participants/total number of contact attempts made
Feasibility - Staff hours per week | End of study (week 48)
  Hours spent providing remote incentives
Feasibility - Adverse effects of incentives | End of study (week 48)
  Unexpected risks/harms of providing incentives as self-reported by participants.
Percentage of participants who are satisfied with the incentive intervention | Enrollment (week 0) and end of study (week 48)
  To assess participant satisfaction with the incentive intervention model. Patient satisfaction, assessed by ACASI survey, will be summarized and tabulated for baseline (week 0) and follow-up (week 48) measurements.
Effect of incentives on missed appointment rate | Enrollment (week 0) and end of study (week 48)
  Descriptive statistics of numbers of missed appointments such as mean, interquartile range and median, during each study phase will be computed and compared
Effect of incentives on STI rates | Enrollment (week 0) and end of study (week 48)
  Descriptive statistics of numbers of STI rates such as mean, interquartile range and median, during each study phase will be computed and compared
Change in biological parameters | At weeks 0, 12, 24, 36 and 48
  To measure the effect of the incentive intervention on HIV viral load and CD4+ count. HIV viral load and CD4+ count measured at week 0, 12, 24, 36 and 48 will be summarized and plotted by descriptive statistics, such as mean and standard deviation. Mixed effects models will be applied to explore the effect of the intervention on HIV viral load and CD4+ count.
Overall cost of incentive intervention | End of study (week 48)
  To determine the overall and per patient cost of the incentive intervention model the accumulated overall and per patient cost till week 48 will be summarized and tabulated.
Association between adherence measures | End of study (week 48)
  To describe associations between adherence measures: Wisepill data, pharmacy pill count, pharmacy prescription pick-up data, medication possession ratio, and self-report. Associations of Wisepill adherence rates with pill count and pick up rates will be described by Pearson or Spearman's correlation coefficients and intraclass correlation coefficients as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Dallas, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols